CLINICAL TRIAL: NCT00059917
Title: Phase I Study of CT-2106 in Patients With Advanced Malignancy
Brief Title: Polyglutamate Camptothecin in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CTI-PGC101; MSKCC-03002; CDR0000298987 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2005-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — polyglutamate camptothecin

INTERVENTIONS:
Drug: polyglutamate camptothecin

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as polyglutamate camptothecin may be able to deliver the drug directly to tumor cells while leaving normal cells undamaged.

PURPOSE: Phase I trial to study the effectiveness of polyglutamate camptothecin in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of polyglutamate camptothecin (CT-2106) in patients with advanced malignancies.
* Determine the tolerability of this drug in these patients.
* Determine the safety of this drug in these patients.
* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.
* Determine the disease response in patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive polyglutamate camptothecin (CT-2106) IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients receive 2 additional courses beyond confirmation of complete response.

Cohorts of 3-6 patients receive escalating doses of CT-2106 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 weeks.

PROJECTED ACCRUAL: A total of 12-48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced malignancy
* No active brain metastases (as indicated by clinical symptoms, cerebral edema, or progressive tumor growth) that have been unstable for at least 8 weeks

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine no greater than 1.5 times ULN
* No history of hemorrhagic cystitis
* No history of microscopic hematuria associated with drug therapy or radiotherapy or of unknown origin

Cardiovascular

* No significant cardiac disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to comply with study schedule and assessments
* No other significant nonmalignant systemic disease
* No active infection
* No other condition that would in the investigator's opinion make the patient an inappropriate study candidate

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 3 prior chemotherapy regimens
* More than 4 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior definitive radiotherapy (except for palliative reasons to sites of nonmeasurable disease, in patients with measurable disease at baseline)
* Concurrent palliative radiotherapy allowed

Surgery

* More than 4 weeks since prior major thoracic or abdominal surgery

Other

* Recovered from prior therapy (except alopecia or stable grade 1 neuropathy)
* More than 4 weeks since prior investigational agents
* No prior myeloablative therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Dupont, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] McNamara MV, Doroshow JH, Dupont J, et al.: Preliminary pharmacokinetics of CT-2106 (polyglutamate camptothecin) in patients with advanced malignancies. [Abstract] J Clin Oncol 22 (Suppl 14): A-2073, 145s, 2004.
- [Result] Springett GM, Takimoto C, McNamara M, et al.: Phase I study of CT-2106 (polyglutamate camptothecin) in patients with advanced malignancies. [Abstract] J Clin Oncol 22 (Suppl 14): A-3127, 226s, 2004.